CLINICAL TRIAL: NCT00458289
Title: Efficacy of Phosphate Binding in Healthy Volunteers: Chewed Versus Crushed Lanthanum Carbonate
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Shire (Industry)
Responsible Party: Principal Investigator, Alan Lau, Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2006-0530
Record Dates: First submitted 2007-04-06; First posted 2007-04-10 (Estimated); Last update posted 2019-12-20 (Actual); Status verified 2019-12

CONDITIONS: Hyperphosphatemia in Chronic Kidney Disease
MeSH Terms: interventions — lanthanum carbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (No Intervention): P-containing meal alone
- 2 (Active Comparator): P-containing meal AND single 1 g oral dose of chewed lanthanum carbonate
  Interventions: Drug: Lanthanum carbonate (chewed vs. crushed)
- 3 (Active Comparator): P-containing meal and single 1 g oral dose of lanthanum carbonate crushed into a fine powder
  Interventions: Drug: Lanthanum carbonate (chewed vs. crushed)

INTERVENTIONS:
Drug: Lanthanum carbonate (chewed vs. crushed) — single 1 g oral dose of lanthanum carbonate either chewed or crushed into a fine powder
  Arms: 2; 3

SUMMARY:
Patients with end-stage renal disease (ESRD) commonly have high concentrations of phosphorous, a mineral, in the blood (hyperphosphatemia). This is a result of their inability to excrete phosphorous by the kidneys. This in turn may result in the development of a condition known as secondary hyperparathyroidism and renal osteodystrophy or bone disease. As such, these patients often receive medications known as phosphate binders such as calcium carbonate or acetate, sevelamer, aluminum hydroxide and lanthanum carbonate to manage and treat hyperphosphatemia.

Lanthanum carbonate is a newly available phosphate binding agent that is effective in the management of hyperphosphatemia and preventing secondary hyperparathyroidism. It works in the gastrointestinal tract by binding to the phosphorus in the diet. ESRD patients taking lanthanum carbonate are counseled to chew the tablets completely before swallowing, with or immediately after meals. However, patients who are intubated or receiving nutrition via feeding tubes are unable to chew the tablets. For these patients, medications are commonly crushed and administered via the tube. Moreover, some patients prefer to crush the tablets and mix it with food instead of chewing. To date, it is not known if crushing the lanthanum carbonate tablets prior to administration and taking it with food would be as effective as chewing them.

The purpose of this study is to compare the efficacy of phosphate binding between chewed and crushed lanthanum carbonate tablets.

ELIGIBILITY:
Inclusion Criteria:

* Men and women at least 18 years of age
* No clinically significant abnormal findings on clinical laboratory evaluation and medical history
* Within 15% of ideal body weight for height and build according to the Metropolitan Life tables5
* Women of child-bearing potential (premenopausal and not surgically sterilized) who have a negative pregnancy test
* Women who are sexually active must be using effective means of contraception

Exclusion Criteria:

* History of dysphagia or swallowing disorders
* Clinically significant illness within 3 months of study enrollment
* Concomitant use of medication that might interact with lanthanum carbonate
* Pregnant or intends to become pregnant within 30 days of completing the study
* Breast feeding
* Alcohol or controlled substance abuse
* Use of an investigational agent within 30 days of study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2007-01; Primary Completion 2008-06 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Serum phosphorous concentration | Hourly from time=0-8 h after administration of meal and drug

CONTACTS AND LOCATIONS:
Overall Officials: Alan H Lau, Pharm.D., Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Dept of Pharmacy Practice, Chicago, Illinois, United States